CLINICAL TRIAL: NCT04264637
Title: A Randomized, Double-Blind, Placebo Controlled, Crossover Study to Evaluate the Onset of Efficacy of Azelastine Hydrochloride 0.15% Nasal Spray in Allergic Rhinitis Sufferers Following Pollen Exposure in an Environmental Exposure Chamber
Brief Title: Study to Find Out How Long it Takes Azelastine Hydrochloride 0.15% Nasal Spray to Relieve Symptoms in Patients Suffering From Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20877
Record Dates: First submitted 2020-02-10; First posted 2020-02-11 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — azelastine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azelastine hydrochloride 0.15% + Placebo (Experimental): Each participant will receive a single dose (two sprays per nostril) of study intervention Azelastine hydrochloride 0.15% and Placebo at treatment period 1 and 2 respectively.
  Interventions: Drug: Azelastine hydrochloride (BAYR9258); Drug: Placebo
- Placebo + Azelastine hydrochloride 0.15% (Experimental): Each participant will receive a single dose (two sprays per nostril) of study intervention Placebo and Azelastine hydrochloride 0.15% at treatment period 1 and 2 respectively.
  Interventions: Drug: Azelastine hydrochloride (BAYR9258); Drug: Placebo

INTERVENTIONS:
Drug: Azelastine hydrochloride (BAYR9258) — Single dose, metered-spray solution, 2 sprays per nostril, 205.5 mcg/spray, intranasal administration.
Drug: Placebo — Single dose of Azelastine hydrochloride-matched placebo, metered-spray solution, 2 sprays per nostril, intranasal administration.

SUMMARY:
In this study researchers want to learn how quickly patients suffering from allergic rhinitis (also known as hay fever) can expect symptom relief after using Azelastine Hydrochloride 0.15% Nasal Spray.

This study plans to enrol about 80 male or female participants in the age of 18 to 65 years suffering from an allergic rhinitis to ragweed pollen for at least 2 years. In a first phase participants will be exposed to ragweed pollen in a special study room to ensure they will be adequately symptomatic when they progress into the treatment phase of the study. In a second phase study participants will be divided in 2 groups. After exposure to ragweed pollen one group will receive Azelastine Hydrochloride 0.15% Nasal Spray and the other group will receive placebo (a nasal spray which does not contain any active drug substance). In the third phase of study the treatment will be switched: participants who received in the previous study Azelastine Hydrochloride 0.15% Nasal Spray will receive the nasal spray without any active drug substance and the other group will receive Azelastine Hydrochloride 0.15% Nasal Spray. During the second and third study phase the researchers will examine thoroughly over 4 hours the change of nasal symptoms such as runny nose, itchy nose, sneezing and nasal congestion after participants received the nasal spray.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male or female volunteers 18 to 65 years of age with selfreported allergic rhinitis to ragweed pollen for at least 2 years prior.
* Documented positive skin prick test response to common ragweed (ambrosia artemisiifolia) pollen; prick with wheal ≥3 mm larger than the diluent response at screening or within the previous 12 months done at the research site.
* Subject is willing to abstain use of any decongestant and/or allergy medications (prescription and over-the-counter), smoking, wearing perfume and alcohol 24 hours prior to the Qualification and Treatment Phases as instructed.
* Subject is willing to stop use of current decongestant and allergy medications at the start of the washout period prior to qualification and during the trial as instructed.
* At the discretion of the investigator, subjects may be considered with self-reported mild intermittent asthma (using ≤2 doses of SABA (short-acting beta agonists) per week) or exercise-induced asthma.
* Female subjects of childbearing potential must: a) be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives); b) abstain from sexual intercourse for at least 1 month prior to screening; or c) participate exclusively in a same sex relationship for at least 1 month prior to screening. In addition, female subjects of childbearing potential must have a negative pregnancy test at Screening and prior to entering the Environmental Exposure Chamber (EEC). Female subjects of non-childbearing potential must be amenorrheic for at least two years or have undergone surgical sterilization (i.e. tubal ligation/occlusion, hysterectomy and/or bilateral oophorectomy).
* At the end of the 4 hour Qualification Phase, the subject's Total Nasal Symptom Score (TNSS) via Electronic Patient Data Acquisition Tablet (ePDAT) must be ≥6 out of a possible of 12 at least twice, with at least one occurring during the last 2 time points to qualify to receive study intervention.
* During Treatment Phases Treatment 1 (T1) and Treatment 2 (T2), subjects are exposed to pollen in EEC for a two hour induction phase. At the end of the two hour symptom induction phase during T1 and T2, subjects meet a minimum threshold total nasal symptom score (TNSS) response of ≥6 out of a possible of 12 at least twice, with at least one occurring during the last 2 time points to qualify to receive study intervention.

Exclusion Criteria:

* Any significant medical condition which, in the judgment of the investigator, is a contraindication to the use of intranasal azelastine hydrochloride (HCl), or might interfere with the trial.
* Subjects with a pre-EEC TNSS ˃3 at T1.
* Subjects with a known allergy to azelastine HCl or any of its inactive ingredients, or with a known contraindication to the use of epinephrine.
* Subjects with a known history of non-allergic rhinitis.
* Subjects with a suspected or known history of anaphylaxis to ragweed allergen.
* Subjects with a suspected or known history of rhinitis medicamentosa.
* In the judgment of the investigator, any respiratory illness or active local infection (e.g., sinusitis) prior to the Qualification Phase that can interfere with the conduct of the study.
* Subjects with a known history of coronary heart disease, ischemic heart disease , high blood pressure, symptomatic prostatic hypertrophy, hepatic insufficienHas a history of immunological disease or malignancy within the past 5 years, with the exception of non-melanoma skin cancer or renal disease.
* Evidence or history of clinically significant (in the judgment of the investigator) hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including hypertension), hepatic, psychiatric, neurologic diseases, or malignancies within the last 5 years.
* Self-reported medical history of tuberculosis, hepatitis or human immunodeficiency virus (HIV).
* Alcoholism or drug abuse within 2 years prior to the Screening Visit or routine consumption of 3 or more alcohol containing beverages per day; Alcohol containing beverages are defined as one beer (5%), one glass of wine (11%) and one shot (40%) hard liquor.
* Self-reported current heavy smokers (>1 pack/25 cigarettes per day).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Total nasal symptom score (TNSS) | 4 hours post dose
  Evaluated by rating the following symptoms (sneezing, runny nose, itchy nose, and nasal congestion) on a scale from 0-3 (0 = None, 1= Mild symptoms, 2 = Moderate symptoms, 3 = Severe symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Hsu SN, Sajjad F, Brigham E, Centofanti R, An R, Couroux P, Ng C. Onset of efficacy of azelastine hydrochloride 0.15% nasal spray for allergic rhinitis in an environmental exposure chamber. Ann Allergy Asthma Immunol. 2024 Dec;133(6):675-681. doi: 10.1016/j.anai.2024.07.020. Epub 2024 Jul 26. PMID 39067509